CLINICAL TRIAL: NCT00532064
Title: Early Detection of Cardiotoxicity During Sunitinib or Sorafenib Chemotherapy Using Cardiac Biomarkers
Brief Title: Cardiac Biomarkers in Early Detection of Cardiotoxicity in Patients Receiving Sunitinib or Sorafenib Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: Terminated per PI's request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0921; NCI-2018-02471 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0921 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection): Patients receive sunitinib malate or sorafenib chemotherapy then undergo blood collection 2 weeks later, and then every 4-6 weeks for up to 6 months to test for troponin I and BNP.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well cardiac biomarkers work in the early detection of cardiotoxicity in patients receiving sunitinib malate or sorafenib chemotherapy. Some chemotherapies are known to cause damage to heart muscle cells, resulting in heart failure. Often, the damage is not detected until heart failure has already occurred. Testing for cardiac biomarkers, such as troponin I and/or T and B-type natriuretic peptide (BNP), may be useful in detecting heart damage earlier than other tests currently performed (such as echocardiogram and electrocardiogram).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if specific biomarkers (troponin I and B-type natriuretic peptide [BNP]) detect cardiotoxicity earlier than standard clinical means in patients receiving sunitinib malate (SU11248) or sorafenib chemotherapy.

SECONDARY OBJECTIVES:

I. To prospectively evaluate the incidence and severity of cardiac toxicity related to sunitinib or sorafenib during chemotherapy.

OUTLINE:

Patients receive sunitinib malate or sorafenib chemotherapy then undergo blood collection 2 weeks later, and then every 4-6 weeks for up to 6 months to test for troponin I and BNP.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18-85 years
* Starting a new course of chemotherapy at MD Anderson Cancer Center that includes sunitinib or sorafenib
* Has a life expectancy of greater than 6 months

Exclusion Criteria:

* Unstable angina within the last 3 months
* Myocardial infarction within the last 3 months
* Left ventricular ejection fraction (LVEF) less than 40%
* Decompensated heart failure (HF) in the last 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDACC Cancer Participants
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2007-09-12 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of each biomarker for detecting cardiotoxicity | Up to 6 months
  Will estimate with exact 95% confidence intervals.
Specificity of each biomarker for detecting cardiotoxicity | Up to 6 months
  Will estimate with exact 95% confidence intervals.

SECONDARY OUTCOMES:
Incidence of cardiotoxicity | Up to 6 months
  Will use the methods of Gooley, et al (1999) to estimate the cumulative incidence of cardiotoxicity while considering deaths from other causes as a competing risk. Will estimate the cumulative incidence of cardiotoxicity while stratifying by common risk factors (one at a time). Will use mixed linear models to model the biomarker levels over time, accounting for the correlation between biomarker levels within patient. Will use logistic regression to model the log odds of cardiotoxicity as a function of common risk factors for cardiotoxicity. Will also include the duration of chemotherapy use and the MD Anderson Symptom Inventory - Heart Failure (MDASI-HF) score as a potential prognostic factor for cardiotoxicity.
MD Anderson Symptom Inventory - Heart Failure (MDASI-HF) score | Up to 6 months
  Will summarize the MD Anderson Symptom Inventory - Heart Failure (MDASI-HF) score over time with descriptive statistics and boxplots.

CONTACTS AND LOCATIONS:
Overall Officials: Elie Mouhayar, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org